CLINICAL TRIAL: NCT03861039
Title: A Phase 3, Long-Term Safety Study of Tirzepatide in Combination With Monotherapy of Oral Antihyperglycemic Medications in Patients With Type 2 Diabetes Mellitus (SURPASS J-combo)
Brief Title: A Long-term Safety Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17078; I8F-JE-GPGP (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 5 mg Tirzepatide (Experimental): 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week. Participant received the following pre-treatment oral antihyperglycemic medication (OAM): Sulfonylurea, biguanide, alpha-glucosidase inhibitor, thiazolidinedione, glinide, or sodium-glucose cotransporter type 2 inhibitor.
  Interventions: Drug: Tirzepatide; Drug: Oral antihyperglycemic medication (OAM)
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once a week. Participant received the following pre-treatment oral antihyperglycemic medication (OAM): Sulfonylurea, biguanide, alpha-glucosidase inhibitor, thiazolidinedione, glinide, or sodium-glucose cotransporter type 2 inhibitor.
  Interventions: Drug: Tirzepatide; Drug: Oral antihyperglycemic medication (OAM)
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once a week. Participant received the following pre-treatment oral antihyperglycemic medication (OAM): Sulfonylurea, biguanide, alpha-glucosidase inhibitor, thiazolidinedione, glinide, or sodium-glucose cotransporter type 2 inhibitor.
  Interventions: Drug: Tirzepatide; Drug: Oral antihyperglycemic medication (OAM)

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
Drug: Oral antihyperglycemic medication (OAM) — Oral antihyperglycemic medication (OAM): Sulfonylurea, biguanide, alpha-glucosidase inhibitor, thiazolidinedione, glinide, or sodium-glucose cotransporter type 2 inhibitor.

SUMMARY:
The purpose of this study is to determine the long-term safety of the study drug tirzepatide in combination with oral antihyperglycemic medications in participants with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Participant must:

* Have been diagnosed with type 2 diabetes mellitus based on the World Health Organization classification before the screening visit.
* Have HbA1c ≥7.0% to <11.0%, as determined by the central laboratory at screening.
* Have been taking sulfonylureas, biguanides, thiazolidinedione, alpha-glucosidase inhibitor, glinides, or sodium-glucose cotransporter type 2 inhibitor monotherapy for at least 3 months before screening and have been on the following dose for at least 8 weeks before screening.
* Have body mass index (BMI) of ≥23 kilograms per meter squared at screening.
* Be of stable weight (±5%) during 3 months preceding screening; and agree to not initiate an intensive diet and/or exercise program during the study with the intent of reducing body weight other than the lifestyle and dietary measures for diabetes treatment.

Exclusion Criteria:

Participant must not:

* Have type 1 diabetes mellitus.
* Have had chronic or acute pancreatitis any time prior to study entry.
* Have proliferative diabetic retinopathy or diabetic maculopathy or nonproliferative diabetic retinopathy requiring immediate or urgent treatment.
* Have disorders associated with slowed emptying of the stomach, or have had any stomach surgeries for the purpose of weight loss.
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or blood alanine transaminase (ALT) enzyme level >3.0 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory. Participants with nonalcoholic fatty liver disease (NAFLD) are eligible for participation in this trial only if there ALT level is ≤3.0 the ULN for the reference range.
* Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months.
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2.
* Have been taking weight loss drugs, including over-the-counter medications during the last 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- Japan (34):
  - Akaicho Clinic, Chiba, Chiba
  - Kashiwa hospital, Kashiwa, Chiba
  - Yuri Ono Clinic, Sapporo, Hokkaido
  - Manda Hospital, Sapporo, Hokkaido
  - Miyanomori Hospital, Sapporo, Hokkaido
  - Ikeda Hospital, Amagasaki, Hyōgo
  - Nakamoto Naika Clinic, Mito, Ibaraki
  - Naka Memorial Clinic, Naka, Ibaraki
  - Ohishi Naika Clinic, Tsuchiura, Ibaraki
  - Takai Naika Clinic, Kamakura, Kanagawa
  - Tsuruma Kaneshiro Diabetes Clinic, Yamato, Kanagawa
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - H.E.C. Science Clinic, Yokohama, Kanagawa
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Otsu City Hospital, Ōtsu, Shiga
  - Wakakusa Clinic, Shimotsuke, Tochigi
  - Seiwa Clinic, Adachi-ku, Tokyo
  - HDC Atlas Clinic, Chiyoda City, Tokyo
  - Asahi Life Foundation Adult Disease Research Center, Chuo-ku, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Tokyo Center Clinic, Chuo-ku, Tokyo
  - Tokyo Clinical Trial Centre Fukuwa Clinic, Chuo-ku, Tokyo
  - Kanno Naika, Mitaka, Tokyo
  - Shinjuku Research Park Clinic, Shinjuku-Ku, Tokyo
  - Futata Tetsuhiro Clinic, Fukuoka
  - Morinaga Ueno Clinic, Kumamoto
  - Jinnouchi Hospital, Kumamoto
  - Saiseikai Noe Hospital, Osaka
  - Kitada Clinic, Osaka
  - Kansai Denryoku Hospital, Osaka
  - Abe Diabetes Clinic, Ōita
  - Shizuoka City Shizuoka Hospital, Shizuoka
  - Suruga Clinic, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Mimura H, Oura T, Chin R, Hirase T, Shimono D. Association Between Early Weight Loss and Metabolic Outcomes with Tirzepatide in Japanese Patients with Type 2 Diabetes: A SURPASS J Post Hoc Analysis. Diabetes Ther. 2025 Sep;16(9):1871-1885. doi: 10.1007/s13300-025-01775-y. Epub 2025 Jul 25. PMID 40711720
- [Derived] Kadowaki T, Chin R, Ozeki A, Imaoka T, Ogawa Y. Safety and efficacy of tirzepatide as an add-on to single oral antihyperglycaemic medication in patients with type 2 diabetes in Japan (SURPASS J-combo): a multicentre, randomised, open-label, parallel-group, phase 3 trial. Lancet Diabetes Endocrinol. 2022 Sep;10(9):634-644. doi: 10.1016/S2213-8587(22)00187-5. Epub 2022 Jul 30. PMID 35914542
- See also: A Long-term Safety Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/2qJ9f49B7nrO6hGapNnDZD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Started | 148 | 147 | 148
Received at Least One Dose of Study Drug | 148 | 147 | 148
Completed | 145 | 139 | 133
Not Completed | 3 | 8 | 15
Not completed — Adverse Event | 2 | 5 | 11
Not completed — Withdrawal by Subject | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Total
Number analyzed (Participants) | 148 | 147 | 148 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (11.0) | 56.9 (11.2) | 56.5 (10.4) | 57.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 44 | 107
  Male | 119 | 113 | 104 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 148 | 147 | 148 | 443
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 148 | 147 | 148 | 443
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 148 | 147 | 148 | 443
Hemoglobin A1c [Mean (Standard Deviation); unit: : Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  : Percentage of HbA1c | 8.53 (1.15) | 8.56 (1.05) | 8.59 (1.09) | 8.56 (1.09)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any AE from this study that results in one of the following outcomes:
  * Death
  * Initial or prolonged inpatient hospitalization
  * A life-threatening experience (that is, immediate risk of dying)
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect.
  * Important medical events that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the patient or may require.
  A summary of all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through Week 52
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 15 mg Tirzepatide: 15 mg tirzepatide administered SC once a week.Participant received the following pre-treatment oral antihyperglycemic medication (OAM): Sulfonylurea, biguanide, alpha-glucosidase inhibitor, thiazolidinedione, glinide, or sodium-glucose cotransporter type 2 inhibitor.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 147 | 148
Participants | 0 | 1 | 1

2. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model for post-baseline measures: Variable = Baseline + oral antihyperglycemic medication (OAM) Group 1 + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 146 | 145
Percentage of HbA1c | -2.57 (0.075) | -2.98 (0.075) | -3.02 (0.077)

3. Secondary Outcome: Percentage of Participants Who Achieve HbA1c <7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 146 | 145
percentage of participants | 92.57 | 97.95 | 96.55

4. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: Fasting serum glucose (FSG) is a test to determine sugar levels in serum sample after an overnight fast. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + OAM Group 1 + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milligram per Deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 146 | 145
milligram per Deciliter (mg/dL) | -58.6 (1.75) | -71.2 (1.75) | -74.4 (1.81)

5. Secondary Outcome: Mean Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Postmeal, Midday Premeal, Midday 2-hour Postmeal, Evening Premeal, Evening 2-hour Postmeal and Bedtime. LS mean was determined by analysis of covariance (ANCOVA) model for endpoint measures: Variable = Baseline + OAM Group 1 + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 136 | 135 | 125
mg/dL | -80.0 (1.91) | -94.1 (1.92) | -96.3 (1.99)

6. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + OAM Group 1 + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 146 | 145
Kilograms (kg) | -3.8 (0.51) | -7.5 (0.51) | -10.2 (0.52)

7. Secondary Outcome: Percentage of Participants Who Achieve Weight Loss of ≥5% From Baseline
Description: Percentage of Participants who Achieve Weight Loss of ≥5% from Baseline
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 146 | 145
percentage of participants | 43.92 | 70.55 | 84.14

8. Secondary Outcome: Change From Baseline in Fasting Insulin
Description: LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement) = log(Baseline) + OAM Group 1 + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: picomol per liter (pmol/L)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 143 | 144 | 134
picomol per liter (pmol/L) | 6.2 (2.68) | -4.8 (2.21) | -7.7 (2.16)

9. Secondary Outcome: Change From Baseline in Fasting C-Peptide
Description: as for outcome 8
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: micrograms/litre (ug/L)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 143 | 144 | 134
micrograms/litre (ug/L) | -0.12 (0.044) | -0.28 (0.040) | -0.34 (0.040)

10. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment B (HOMA-2B) (Insulin)
Description: The HOMA2 is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state pancreatic beta cell function (%B) and to estimate insulin sensitivity (%S) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. The change from baseline for fasting insulin concentrations are presented as insulin secretion (HOMA2-%B) and insulin sensitivity (HOMA2-%S).
  LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement) = log(Baseline) + OAM Group 1 + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA-2B
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 139 | 135 | 128
percentage of HOMA-2B | 39.7 (2.16) | 44.9 (2.40) | 49.2 (2.60)

11. Secondary Outcome: Change From Baseline in HOMA-2S (Insulin)
Description: as for outcome 10
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of HOMA-2S
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 139 | 135 | 128
Percentage of HOMA-2S | -0.1 (3.37) | 16.7 (4.23) | 24.1 (4.66)

12. Secondary Outcome: Number of Participants With Hypoglycemia Incidence and Rate With Blood Glucose <54 mg/dL or Severe Hypoglycemia, Exclude Hypoglycemic Events Occurring After Initiation of a New Antihyperglycemic Therapy
Description: The hypoglycemia events were defined by participant reported events with blood glucose <54mg/dL (<3.0 mmol/L) or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Baseline through Week 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg Tirzepatide: 10 mg tirzepatide administered SC once a week.Participant received the following pre-treatment oral antihyperglycemic medication (OAM): Sulfonylurea, biguanide, alpha-glucosidase inhibitor, thiazolidinedione, glinide, or sodium-glucose cotransporter type 2 inhibitor.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 147 | 148
Participants | 1 | 1 | 3

13. Secondary Outcome: Number of Participants With Anti-Tirzepatide Antibodies
Description: Number of Participants with Anti-Tirzepatide Antibodies
Time Frame: Baseline through Week 52
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 148 | 147 | 148
Participants | 87 | 82 | 88

ADVERSE EVENTS:
Time Frame: Baseline through Week 56
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- 5 mg Tirzepatide: 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.Participant received the following pre-treatment oral antihyperglycemic medication (OAM): Sulfonylurea, biguanide, alpha-glucosidase inhibitor, thiazolidinedione, glinide, or sodium-glucose cotransporter type 2 inhibitor.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/147 | 0/148
Serious Adverse Events (participants affected / at risk) | 2/148 | 11/147 | 11/148
Other Adverse Events (participants affected / at risk) | 109/148 | 108/147 | 124/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=148) | 10 mg Tirzepatide (N=147) | 15 mg Tirzepatide (N=148)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intra-cerebral aneurysm operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=148) | 10 mg Tirzepatide (N=147) | 15 mg Tirzepatide (N=148)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Corneal leukoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 9 (10) | 7 (9) | 8 (10)
Abdominal distension (Gastrointestinal disorders) | 5 (6) | 6 (7) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 4 (4) | 5 (5)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 12 (12) | 20 (21) | 22 (24)
Dental caries (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (24) | 20 (40) | 20 (28)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 11 (19) | 5 (6)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 6 (6) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (60) | 20 (35) | 40 (51)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 11 (13) | 15 (23)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (4) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (4)
Fatigue (General disorders) | 2 (2) | 2 (2) | 3 (4)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Injection site reaction (General disorders) | 4 (7) | 3 (25) | 4 (72)
Malaise (General disorders) | 2 (2) | 3 (4) | 6 (6)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Fatty liver alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Adenoviral conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (6)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 7 (9) | 5 (5) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 1 (1) | 2 (2)
Nasal vestibulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 28 (34) | 20 (26) | 27 (37)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Rhinitis (Infections and infestations) | 3 (4) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/29 (0) | 2/34 (2) | 1/44 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (3) | 2 (3) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 2 (3) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood calcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 2 (3) | 1 (1) | 1 (1)
Electrocardiogram st segment depression (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter test positive (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Lipase increased (Investigations) | 4 (5) | 4 (4) | 9 (9)
Occult blood (Investigations) | 0 (0) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Salmonella test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 8 (8) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 15 (18) | 18 (19)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Hypercalcitoninaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/29 (0) | 0/34 (0) | 1/44 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 8 (8)
Dizziness postural (Nervous system disorders) | 0 (0) | 3 (6) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 2 (2) | 1 (1) | 4 (4)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/119 (0) | 1/113 (1) | 0/104 (0)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0/29 (0) | 1/34 (1) | 0/44 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0/29 (0) | 1/34 (1) | 0/44 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 3 (3)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Skin lesion removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ureteric calculus removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Urethral stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT03861039/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT03861039/SAP_001.pdf